CLINICAL TRIAL: NCT06984601
Title: RELIEF Study: Resolving Fissures With Lateral Internal Sphincterotomy - Evaluating Function and Quality of Life: A National, Prospective Cohort Study
Brief Title: RELIEF Study: Resolving Fissures With Lateral Internal Sphincterotomy
Acronym: RELIEF
Status: Not yet recruiting | Type: Observational
Sponsor: Turkish Society of Colon and Rectal Surgery (Other)
Responsible Party: Sponsor
Other Study IDs: 187
Record Dates: First submitted 2025-04-30; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-04

CONDITIONS: Chronic Anal Fissure
Keywords: Chronic anal fissure; Lateral internal sphincterotomy; Fecal incontinence
MeSH Terms: conditions — Fecal Incontinence | interventions — Lateral Internal Sphincterotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tailored LIS: Participants undergoing tailored lateral internal sphincterotomy, with sphincter division based on spasm severity or fissure characteristics
  Interventions: Procedure: Lateral Internal Sphincterotomy (LIS)
- Classical LIS: Participants undergoing traditional sphincterotomy, with incision to the fissure apex or a fixed anatomical point
  Interventions: Procedure: Lateral Internal Sphincterotomy (LIS)

INTERVENTIONS:
Procedure: Lateral Internal Sphincterotomy (LIS) — This is a routinely performed surgical procedure for chronic anal fissure. The study is observational and does not assign this procedure to participants.

SUMMARY:
The goal of this observational study is to learn how a common surgery called lateral internal sphincterotomy (LIS) affects people with chronic anal fissures, a painful tear near the anus. The study will look at whether this surgery helps lower problems like pain and incontinence, and how it affects quality of life and mental health.

The main questions the study aims to answer are:

Does LIS surgery lower the rate of incontinence one year after surgery? Does it improve quality of life, reduce pain, and increase patient satisfaction?

Participants will:

Have surgery for chronic anal fissure called LIS. Complete short surveys about pain and mental health at 1 week, 3 months, and 12 months.

Answer questions about bowel function, incontinence and daily life at 3 and 12 months.

Researchers will follow about 300 adults at hospitals across the Turkey. This study will help improve future treatment decisions and make surgery safer and more effective.

DETAILED DESCRIPTION:
Chronic anal fissure is a common anorectal condition that can significantly affect daily life due to pain and difficulty with bowel movements. Lateral internal sphincterotomy (LIS) is a widely used surgical treatment for fissures that do not improve with medical therapy. While LIS is highly effective in promoting healing, it may lead to complications such as fecal incontinence, which can negatively affect quality of life.

The RELIEF Study is a prospective, multicenter cohort study conducted across several hospitals in Turkey. The aim is to evaluate the long-term effects of LIS on bowel control, postoperative pain, patient satisfaction, and mental health. Participants will be followed for 12 months after surgery. Data will be collected using a secure electronic data capture system (REDCap) to ensure standardization and data quality.

Approximately 300 adult participants will be enrolled. Researchers will examine different surgical approaches to LIS, including tailored techniques (based on fissure location or sphincter tone) and classical methods (such as sphincterotomy to the fissure apex). By comparing outcomes across these techniques, the study will help identify safer and more effective strategies.

Validated tools, including incontinence scores, pain scales, and quality of life questionnaires, will be used to measure outcomes. The findings are expected to inform clinical practice and contribute to the development of evidence-based guidelines for the treatment of chronic anal fissures.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Diagnosed with chronic anal fissure (symptoms lasting more than 6 weeks)
* Decision for lateral internal sphincterotomy (LIS) made by the treating physician
* Able to understand and complete study-related questionnaires

Exclusion Criteria:

* Presence of other anorectal or rectal diseases (e.g., fistula, abscess, inflammatory bowel disease)
* History of prior anal surgery or pelvic radiation
* Inability to comprehend study-related forms or provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged 18 years or older diagnosed with chronic anal fissure who are undergoing lateral internal sphincterotomy (LIS) as part of routine clinical care. Participants will be recruited from multiple surgical centers across Turkey. The study includes both male and female patients with no upper age limit.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with a clinically significant change in fecal incontinence | Baseline, 12 months postoperatively
  A clinically significant improvement is defined as a reduction of ≥2 points in the Cleveland Clinic Incontinence Score (Wexner Score), which ranges from 0 (perfect continence) to 20 (complete incontinence). Higher scores indicate worse fecal incontinence. The proportion of patients achieving this threshold will be calculated at 12 months postoperatively.

SECONDARY OUTCOMES:
Fecal Incontinence Quality of Life (FIQoL) Scale Score | Baseline, 3 - 12 months after surgery
  The Fecal Incontinence Quality of Life (FIQoL) scale is a 29-item patient-reported questionnaire that assesses quality of life in patients with fecal incontinence. It consists of four subscales (Lifestyle, Coping/Behavior, Depression/Self-Perception, and Embarrassment). Each item is scored from 1 to 4, with subscale scores calculated as the average of the corresponding item scores. Possible scores range from 1 (minimum) to 4 (maximum), with higher scores indicating better quality of life.
Short Form-36 (SF-36) Health Survey Score | Baseline, 3 - 12 months after surgery
  The Short Form-36 (SF-36) Health Survey is a validated 36-item questionnaire assessing health-related quality of life across 8 domains: Physical Functioning, Role Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role Emotional, and Mental Health. Each domain is scored on a scale from 0 to 100, with higher scores indicating better health status. Composite summary scores (Physical and Mental Component Summary) may also be calculated.
Change in disease-specific quality of life measured by the Hemo-Fiss-QoL questionnaire | Baseline, 3 - 12 months after surgery
  The Hemo-Fiss-QoL is a validated disease-specific tool for assessing quality of life in patients with hemorrhoids or anal fissure. Total scores range from 0 to 100, with higher scores indicating worse quality of life.
Change in Anxiety and Depression Scores (HADS) | 7-10 days, 3 months, 12 months
  Anxiety will be assessed using the Hospital Anxiety and Depression Scale - Anxiety Subscale (HADS-A). This subscale includes 7 items, each scored from 0 to 3, yielding a total score from 0 (no anxiety) to 21 (severe anxiety). Higher scores indicate worse anxiety symptoms.
Change in Pain Scores Using Visual Analog Scale (VAS) | 7-10 days, 3 months, 12 months
  Postoperative pain will be assessed using the Visual Analog Scale (VAS), a 10-point scale ranging from 0 (no pain) to 10 (worst imaginable pain). Patients will self-report their pain intensity. Higher scores indicate worse pain.
Patient Satisfaction Score | 12 months after surgery
  Patient satisfaction with the surgical outcome will be assessed using a self-reported 5-point Likert scale, where:
  1 = Very Dissatisfied, 2 = Dissatisfied, 3 = Neutral, 4 = Satisfied, 5 = Very Satisfied Higher scores indicate greater satisfaction with treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Sezai Leventoğlu, Proffesor, Study Chair — Gazi University

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared upon reasonable request. Data will be anonymized and made available to qualified researchers after approval by the study committee.
Supporting Information: Study Protocol, ICF